CLINICAL TRIAL: NCT04482478
Title: A 12 Week, Randomized, Double-blind, Placebo-Controlled Clinical Trial for the Evaluation of the Efficacy and Safety of EDL on Dyspepsia
Brief Title: Clinical Trial for the Evaluation of the Efficacy and Safety of EDL on Dyspepsia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Bundang Hospital (Other)
Responsible Party: Principal Investigator, Nayoung Kim, Professor, Seoul National University Bundang Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NOVAKM_EDL
Record Dates: First submitted 2020-07-14; First posted 2020-07-22 (Actual); Last update posted 2024-11-29 (Actual); Status verified 2024-11

CONDITIONS: Functional Dyspepsia
Keywords: Functional Dyspepsia; GSRS

STUDY DESIGN:
Intervention Model Description: Subjects are randomly assigned to either the test group or the control group according to the registered order. Subjects take investigational product or placebo for 12 weeks.
  Investigational product (EDL): once a day, 2 tablets orally intake (Extract of Dolichos lablab Linne 715 mg/day) Placebo: consumed in the same way as the investigational product
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- EDL(Extract of Dolichos lablab Linne) (Experimental): The randomly assigned target was given a Extract of Dolichos lablab Linne (EDL) 715 mg/day for 12 weeks.
  Interventions: Dietary Supplement: Extract of Dolichos lablab Linne (EDL)
- Placebo comparator (Placebo Comparator): The randomly assigned target was given a placebo for 12 weeks.
  Interventions: Other: Placebo oral tablet

INTERVENTIONS:
Dietary Supplement: Extract of Dolichos lablab Linne (EDL) — Investigational product (EDL): once a day, 2 tablets orally intake (Extract of Dolichos lablab Linne 715 mg/day)
  Arms: EDL(Extract of Dolichos lablab Linne)
Other: Placebo oral tablet — Placebo: consumed in the same way as the investigational product
  Arms: Placebo comparator

SUMMARY:
This clinical trial was designed to evaluate the functional and safety effects on dyspeptic symptoms compared to the placebo when ingested with EDL (Extract of Dolichos lablab Linne) in adults who complain of dyspeptic symptoms.

DETAILED DESCRIPTION:
Dyspepsia is a common disease and accounts for about 5% of all patients visiting primary care. Of these, about 70~90% of dyspeptic patients who visit the tertiary medical institution have functional digestion, considering that about 8~20% of dyspeptic patients who are referred from the primary medical institution to the tertiary medical institution are found. It is estimated to be bad. Functional dyspepsia is not life-threatening, but its symptoms persist throughout life and are not easily cured, which can limit social life and reduce the quality of life.

Therefore, this clinical trial was designed to evaluate the functional and safety effects on dyspeptic symptoms compared to the placebo when ingested with EDL (Extract of Dolichos lablab Linne) in adults who complain of dyspeptic symptoms.

ELIGIBILITY:
Inclusion Criteria:

1. Those over the age of 19
2. Those diagnosed with functional dyspepsia (Rome IV*)

   * One or more of the following symptoms are diagnosed when there is no organic cause in the test including the upper gastrointestinal endoscopy(if symptoms begin 6 months prior to Visit 1, and the symptoms are present in the past 3 months).
   * Othersome postprandial fullness
   * Unpleasant early satiation
   * Unpleasant epigastric pain
   * Unpleasant epigastric burning
3. A person who has 4 or more of the 10 symptoms in the GIS (Gastrointestinal Symptom) questionnaire and has a total score of 12 or more (5-point Likert scale)
4. When there is no organic disease in the gastroscopy performed at Visit 1 (however, it can be replaced by the test results within 3 months from Visit 1)
5. A person who consented to participate in this clinical trial and signed a Informed consent form before the trail began.

Exclusion Criteria:

1. Persons who are currently being treated with severe cardiovascular system, immune system, respiratory system, hepatobiliary system, kidney and urinary system, nervous system, musculoskeletal system, mental, infectious diseases, and malignant tumors (however, considering the condition of the subjects, subjects can participate in the test according to investigator's judgment.)
2. Persons with a history of peptic ulcer and reflux esophagitis within 6 months of Visit 1
3. Those who have gastrointestinal surgery (except appendectomy and hemorrhoidectomy)
4. Persons with a history of malignancy of the digestive system
5. Those who have taken H2 receptor blockers, anticholinergic agents (muscarinic receptor antagonists), gastrin receptor antagonists, prostaglandin preparations, proton pump inhibitors, gastric mucosal protective agents, other drugs intended to treat gastritis, gastric health-related health functional food within 2 weeks of Visit 1
6. Those who need to constantly take medications that can cause gastritis, such as adrenal cortical hormones, nonsteroidal anti-inflammatory drugs, and aspirin during the human application test {However, low-dose aspirin for cardiovascular disease prevention (100 mg/day or less) permit}
7. In the Drinking Habit Questionnaire, those who had an average alcohol intake of 14 units or more for men and or more 7 units for women per week for the past month.
8. Uncontrolled hypertension persons (systolic blood pressure of 160 mmHg or higher, or diastolic blood pressure of 100 mmHg or higher, measurement criteria after 10 minutes of stability in human subjects)
9. Persons with uncontrolled diabetes (fasting blood sugar is over 180 mg/dL)
10. Those whose Creatinine is more than twice the normal upper limit of the study institution
11. Those whose AST(GOT) or ALT(GPT) is more than 3 times the normal upper limit of the study institution
12. Persons who are sensitive or allergic to investigational product for this clinical trial
13. Pregnant, lactating or planning to become pregnant within 3 months
14. Those who participated in other clinical trials within 3 months of Visit 1 or plan to participate in other clinical trials after the start of this clinical trials.
15. A person who determines that the Investigator is inappropriate for clinical trials
16. Employee of Department of Digestive Internal Medicine, Seoul National University Bundang Hospital

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-07-01 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
GSRS(Gastrointestinal Symptom Rating Scale) Stomach symptom score | 12 weeks
  GSRS (Gastrointestinal Symptom Rating Scale) Stomach symptom score change after 12 weeks of administration, compared to Baseline.
  * the unabbreviated scale title: Gastrointestinal Symptom Rating Scale
  * the minimum and maximum values: 0, 24
  * higher scores mean a worse outcome.

SECONDARY OUTCOMES:
GSRS(Gastrointestinal Symptom Rating Scale) Stomach symptom score | 6 weeks
  GSRS (Gastrointestinal Symptom Rating Scale) Stomach symptom score change after 6 weeks of administration, compared to Baseline.
  * the unabbreviated scale title: Gastrointestinal Symptom Rating Scale
  * the minimum and maximum values: 0, 24
  * higher scores mean a worse outcome.
GSRS(Gastrointestinal Symptom Rating Scale) Total score | 6 weeks, 12 weeks
  GSRS (Gastrointestinal Symptom Rating Scale) Total score change after 6 weeks, 12 weeks of administration, compared to Baseline.
  * the unabbreviated scale title: Gastrointestinal Symptom Rating Scale
  * the minimum and maximum values: 0, 45
  * higher scores mean a worse outcome.
GIS(Gastrointestinal Symptom) | 6 weeks, 12 weeks
  GIS(Gastrointestinal Symptom) score change after 6 weeks, 12 weeks of administration, compared to Baseline.
  * the unabbreviated scale title: Gastrointestinal Symptom
  * the minimum and maximum values: 0, 40
  * higher scores mean a worse outcome.
FD-QoL(Functional Dyspepsia-Related Quality of Life) | 12 weeks
  FD-QoL(Functional Dyspepsia-Related Quality of Life) score change after 12 weeks of administration, compared to Baseline.
  * the unabbreviated scale title: Functional Dyspepsia-Related Quality of Life
  * the minimum and maximum values: 0, 84
  * higher scores mean a worse outcome.
ESR(Erythrocyte Sedimentation Rate) | 6 weeks, 12 weeks
  ESR(Erythrocyte Sedimentation Rate) change after 6 weeks, 12 weeks of administration, compared to Baseline.
CRP(C-Reactive Protein) | 6 weeks, 12 weeks
  CRP(C-Reactive Protein) change after 6 weeks, 12 weeks of administration, compared to Baseline.
IFN-γ(Interferon) | 12 weeks
  IFN-γ(Interferon) change after 12 weeks of administration, compared to Baseline.
TNF-α(Tumor necrosis factors) | 12 weeks
  TNF-α(Tumor necrosis factors) change after 12 weeks of administration, compared to Baseline.
8-OhdG(8-Oxo-2'-deoxyguanosine) | 12 weeks
  8-OhdG(8-Oxo-2'-deoxyguanosine) change after 12 weeks of administration, compared to Baseline.
TAS(total antioxidnat status) | 12 weeks
  TAS(total antioxidnat status) change after 12 weeks of administration, compared to Baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Nayoung Kim, M.D., Ph. D., Principal Investigator — Seoul National University Bundang Hospital
Locations (1):
- Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: No